CLINICAL TRIAL: NCT01398501
Title: Phase I Trial of Sorafenib Maintenance Therapy for Patients With FLT3-ITD AML After Allogeneic Stem Cell Transplantation
Brief Title: Sorafenib Maintenance Therapy for Patients With AML After Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-114
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; FLT3-ITD; Stem cell transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post-SCT Sorafenib (Experimental): Sorafenib will be given as maintenance therapy after allo HCT to patients with FLT3-ITD AML.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Oral, 200 to 400 mg QD or BID
  Other Names: BAY 43-9006

SUMMARY:
Sorfenib works by slowing the spread of cancer cells. It has been used in other studies for patients with AML with the FLT3-ITD mutation and information from these studies suggests that sorafenib may help to control leukemia. The purpose of this study is to find the highest dose of sorafenib for maintenance therapy that can be safely used in participants with AML who have undergone allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Subjects will taken sorafenib orally either once or twice daily. Subjects will come to the Bone Marrow Transplant Clinic 3 times (on Day 8, 15, and 30) during the first month of treatment. After the first month, they will be seen every month for 3 months and then at 9 at 6 and 9 months. Subjects will have a physical exam and be asked questions regarding general health and specific questions about any problems they might be having and any medications they are taking.

Subjects will have standard blood tests every month for 12 months to check liver and kidney function and complete blood count.

Subjects will have research blood tests on Days 8, 15 and 30 during the first month of treatment.

Subjects will have a bone marrow biopsy after 3 months and 12 months of treatment.

Subjects will receive treatment for up to 12 months and be followed for 1 year after completing the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with AML with the FLT3-ITD mutation who have undergone allogeneic HSCT
* Peripheral blood chimerism studies showing >/= 70% of all cells are of donor origin
* Adequate hematologic and hepatic function
* ECOG performance status 0-2
* Able to swallow whole pills

Exclusion Criteria:

* Evidence of relapsed/recurrent/residual disease as assessed by bone marrow aspirate and biopsy performed between days 30-60 after HSCT
* Active acute graft vs host disease requiring an equivalent dose of > 0.5 mg/kg/day of prednisone or equivalent or those patients which necessitated the addition of another agent for the treatment of GVHD beyond corticosteroids
* Ongoing uncontrolled infection
* Cardiac disease: congestive heart failure > class II NYHA, unstable angina or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension
* Known HIV infection or chronic hepatitis B or C
* Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE v 4.0 Grade 2 within 4 weeks of starting study drug
* Any other hemorrhage/bleeding event > CTCAE v. 4.0 Grade 3 within 4 weeks of starting study drug
* Serious non-healing wound, non-healing ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery or significant traumatic injury within 4 weeks of starting study drug
* Use of St. John's Wort or rifampin (rifampicin)
* Known or suspected allergy to sorafenib
* Pregnant or breast-feeding
* Receiving any other investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 3 years
  To define the maximum tolerated dose (MTD) of maintenance sorafenib after allogeneic HSCT

SECONDARY OUTCOMES:
Median number of days sorafenib tolerated | 3 years
  Define the median number of days of sorafenib tolerated prior to dose-limiting toxicity or disease relapse
Rate of serious infections | 3 years
  Rate of serious infections (bacterial, viral, fungal, or other) after starting sorafenib
Rate of acute GVHD | 3 years
  Rate of grades II-IV acute graft-vs-host disease (GVHD) after starting sorafenib
Rate of chronic GVHD | 3 years
  Rates of significant chronic GVHD after starting sorafenib
Survival | 3 years
  1-year and 2-year progression-free and overall survival after HSCT
Impact of sorafenib on bone marrow and serum levels of FLT3-ITD quantitative PCR | 3 years
  To assess the impact of sorafenib on quantitative bone marrow and serum levels of FLT3-ITD DNA in patients (as measured by PCR) with FLT3-ITD AML after allogeneic SCT

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Chen YB, Li S, Lane AA, Connolly C, Del Rio C, Valles B, Curtis M, Ballen K, Cutler C, Dey BR, El-Jawahri A, Fathi AT, Ho VT, Joyce A, McAfee S, Rudek M, Rajkhowa T, Verselis S, Antin JH, Spitzer TR, Levis M, Soiffer R. Phase I trial of maintenance sorafenib after allogeneic hematopoietic stem cell transplantation for fms-like tyrosine kinase 3 internal tandem duplication acute myeloid leukemia. Biol Blood Marrow Transplant. 2014 Dec;20(12):2042-8. doi: 10.1016/j.bbmt.2014.09.007. Epub 2014 Sep 17. PMID 25239228